CLINICAL TRIAL: NCT07035938
Title: An Observational, Bidirectional Cohort Study to Evaluate T-cell Developmental Status in Patients With Malignant Hematological Tumors
Brief Title: T-cell Developmental Status in Patients With Malignant Hematological Tumors
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, Zhijuan Lin, Principal Investigator, The First Affiliated Hospital of Xiamen University
Other Study IDs: XMDYYYXYK-0616
Record Dates: First submitted 2025-06-16; First posted 2025-06-25 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- B-cell lymphoma: Patients with newly diagnosed or relapsed B-cell lymphoma
  Interventions: Other: observational study
- Multiple myeloma: Patients with newly diagnosed or relapsed multiple myeloma
  Interventions: Other: observational study
- HC: Healthy controls
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — observational study

SUMMARY:
To evaluate the immune status and prognosis of patients with malignant hematological tumors, thereby guiding clinical therapeutic strategies.

DETAILED DESCRIPTION:
Primary Objective:

To evaluate the immune status and prognosis of patients with newly diagnosed or relapsed B-cell lymphoma and multiple myeloma by dynamically monitoring peripheral blood thymus seeding progenitors (TSP), recent thymic emigrants (RTE), T-cell receptor rearrangement excision circles (TREC), naive T-cells, and developmental/functional T-cell subsets before and after treatment, thereby guiding clinical therapeutic strategies.

Secondary Objective:

To monitor remission rates, survival outcomes, and infection rates in patients with hematological malignancies, and to explore their association with dynamic changes in developmental/functional T-cell subsets.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years; both genders included; expected survival > 3 months;
2. Cohort 1: Patients with newly diagnosed or relapsed B-cell lymphoma confirmed by histopathology, bone marrow pathology, flow cytometry, morphology, and genetic testing; Cohort 2: Patients with newly diagnosed or relapsed multiple myeloma confirmed by the same methods; Cohort 3: Healthy volunteers;
3. Able to understand and voluntarily sign the informed consent form.

Exclusion Criteria:

1. Significant pulmonary disease:

   Chronic obstructive pulmonary disease (COPD) with forced expiratory volume in 1 second (FEV1) <50% of predicted normal value. Note: Suspected COPD cases require FEV1 testing; subjects with FEV1 <50% of predicted must be excluded.

   Moderate/severe persistent asthma within the past 2 years, or currently uncontrolled asthma of any severity. (Note: Controlled intermittent or mild persistent asthma is permitted.)
2. Symptomatic congestive heart failure (NYHA Class II-IV), symptomatic/uncontrolled arrhythmias, congenital long QT syndrome, or corrected QT interval (QTc) >500 ms (Fridericia formula) at screening.
3. History of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, drug-related pneumonitis, or severely impaired lung function.
4. HIV infection (positive HIV-1/2 antibodies) or known syphilis infection.
5. Unhealed wounds, fractures, gastroduodenal ulcers, persistent fecal occult blood positivity, ulcerative colitis, or other conditions at risk of gastrointestinal bleeding/perforation (as determined by the investigator).
6. Severe neurological/psychiatric disorders, immunodeficiency, hepatitis/cirrhosis, or other conditions deemed unsuitable for study participation by the investigator.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Cohort 1: 25 patients with newly diagnosed or relapsed B-cell lymphoma; Cohort 2: 25 patients with newly diagnosed or relapsed multiple myeloma; Cohort 3: 25 healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-06-22 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentages of TSP/RTE, TREC, and mature T-cell subsets，% | Up to 36 months
  Dynamic changes in peripheral blood TSP/RTE, TREC, and mature T-cell subsets before treatment initiation, before the 2nd, 3rd, and 5th treatment cycles

CONTACTS AND LOCATIONS:
Locations (1):
- Zhijuan Lin, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No